CLINICAL TRIAL: NCT03011502
Title: InterventiOnal Study of Bone and Joint Infections Related Gut dysbiosIS
Acronym: OSIRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MPBJI01
Record Dates: First submitted 2016-12-27; First posted 2017-01-05 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-11

CONDITIONS: Bone and Joint Infection
MeSH Terms: interventions — Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Other: Biological samples collection of blood and feces

INTERVENTIONS:
Other: Biological samples collection of blood and feces

SUMMARY:
Gut dysbiosis is an intestinal disorder that is characterized by accumulation of microbiota imbalance, host-microbiota crosstalk dysfunction and inflammation.

As part of its clinical development, MaaT (Microbiota as a Therapy) Pharma is particularly interested in patients with Bone and Joint Infections (BJI). These patients are treated with antibiotics having significant consequences on their intestinal flora, causing intestinal discomfort, which can be manifested by diarrhea.

MaaT Pharma wishes to carry out a clinical study, OSIRIS, in collaboration with Prof. Tristan Ferry, member and coordinator of CRIOAc (Centre de Référence des Infections Ostéo-Articulaires Complexes) Lyon, Center of Reference of Bone and Joint Infections (BJI). The objective of this study is to follow patients with treated BJI in order to characterize intestinal dysbiosis and the future relevance of an autologous Fecal Microbiota Transplantation (aFMT) intervention.

To do this, patients will be monitored according to the current CRIOAc recommendations, with the aim of taking biological samples from patients at the same time as scheduled visits, routine monitoring patients. Only one additional consultation will be carried out 15 days after stopping the antibiotics in order to better evaluate the dysbiosis evolution.

Thus biological samples (blood, stool, nasal, rectal) will be taken during the follow-up consultations over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Consenting subjects with BJI (native or material related BJI) at participating sites who are being treated with antibiotics as part of their standard treatment procedure will be enrolled
* The subject is willing, able to understand and comply to the protocol requirement
* More than 18-years-old
* Subject is suspected for implanted or native BJI and is eligible for antibiotics treatment
* Subject signed Inform Consent Form

Exclusion Criteria:

* Pregnancy
* Severe disease with a life expectancy < 3 months
* Antibiotherapy in the 14 days before inclusion in the study
* Patient non-affiliated to health care system
* Patient under the power of law
* Guardianship, curators patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
Evolution of intensity and frequency of Diarrheic Symptoms | From baseline, up to 15 days after antibiotherapy treatment stop (Week 8 to week 14)
  Assessment of the evolution of intensity and frequency of Diarrheic Symptoms from baseline, during antibiotic treatment (W2), at the end of treatment (W6-12) and 15 days after antibiotherapy treatment stop (W8-14)

SECONDARY OUTCOMES:
Characterization of the gut dysbiosis and its prevalence in patients with BJI and under antibiotic treatment : measured by NGS (Next-Generation Sequencing) method | Between baseline, after antibiotherapy treatment stop (Week 8-14) and the end of the follow-up (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, MD, PhD, Principal Investigator — Hôpitaux civils de Lyon
Locations (5):
- France (5):
  - CHU Bordeaux, Bordeaux
  - HCL Croix-Rousse, Lyon
  - CHU de Nantes, Nantes
  - GH Diaconesses-Croix Saint Simon, Paris
  - CH Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: Yes